

## Statistical Analysis Plan

Title of Study: Can an adjustable compression garment replace compression bandaging in the treatment of patients with Breast Cancer related upper limb Lymphoedema? A pilot study

Document creation date: March 26th 2020

NCT number [not yet assigned]

Identifiers: [NCT ID not yet assigned]



## Statistical Analysis Plan

- 1. Effect of treatment on primary outcome measure (limb volume measured by circumferential measurements and truncated cone formula) will be determined by using Paired T tests to compare before and after data in both groups.
- 2. SF 36 quality of life analysis An unpaired t-test will be used to compare differences between groups for total scores and also for the subsections of the SF 36.